CLINICAL TRIAL: NCT06772896
Title: Evaluating the Effect of Questionnaire Context on the Reporting of Somatic Items in the 8-item Patient Health Questionnaire Among People With Systemic Sclerosis: A Scleroderma Patient-centered Intervention Network (SPIN) Study
Brief Title: Evaluating the Effect of Questionnaire Context on the Reporting of Somatic Items Among People With Systemic Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Davis Institute (Other)
Responsible Party: Principal Investigator, Brett D Thombs, Senior Investigator, Lady Davis Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2025-PHQ
Record Dates: First submitted 2025-01-07; First posted 2025-01-14 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-01

CONDITIONS: Scleroderma; Systemic Sclerosis (SSc); Scleroderma (Limited and Diffuse)
Keywords: Scleroderma; Systemic Sclerosis; Depression; Patient-reported outcome measure; PROM; Item order
MeSH Terms: conditions — Scleroderma, Diffuse; Scleroderma, Systemic; Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Reordered items (Experimental): Participants will receive a routine assessment protocol in which the 3 PHQ-8 somatic items will be presented separately from and prior to the 5 psychological items, without any indication they are part of a depression symptom questionnaire. PHQ-8 psychological items will be presented after the somatic items and with at least 1 measure separating them in the routine assessment protocol. With the exception of these 2 rules, all measures included in the routine assessment will appear in a random order for each SPIN Cohort participant.
  Interventions: Other: Reordered PHQ-8
- Original item order (No Intervention): Participants will complete the standard version of the PHQ-8 which includes both somatic and psychological items, presented in a random order among other measures of the routine assessment protocol. The title of the PHQ-8 will not be included and participants will only see the 8 items presented on a single page in their standard order.

INTERVENTIONS:
Other: Reordered PHQ-8 — Participants will be administered the PHQ-8 somatic items separately from the psychological items, outside the context of a depression questionnaire.
  Arms: Reordered items

SUMMARY:
There is concern that self-reported depression questionnaires that contain items assessing somatic symptoms may result in biased scores in people with a chronic disease due to symptoms that overlap with their physical disease. However, it has been shown in previous studies that biases associated with somatic items do not affect total depression scores. The reason for this is still unclear but could be associated with the context in which these items are presented.

The goal of this experiment is to learn whether the way people with systemic sclerosis answer somatic items on a depression questionnaire is influenced by the fact that they are aware they are being assessed for depressive symptoms.

The main question it aims to answer is: Do people with systemic sclerosis score somatic items differently when they are administered outside the context of a depression questionnaire? Participants will be randomly assigned to complete the 8-item Patient Health Questionnaire as part of their routine cohort assessments either with the items in their standard order or with somatic items presented first and separately from psychological items.

DETAILED DESCRIPTION:
* BACKGROUND Most self-report depression symptom questionnaires include both psychological and somatic symptom items. The 9-item Patient Health Questionnaire (PHQ-9) and its 8-item version (PHQ-8) are commonly used depression assessment measures and include items that reflect the psychological and somatic symptoms of depression listed in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5). However, there is concern that scores obtained using such questionnaires may be inflated in people with chronic illness due to the overlap of somatic symptoms related to depression and those stemming from their physical illness. In contrast to what might be expected, existing research suggests that having a medical illness or the severity of a respondent's medical illness are not associated with higher scores on somatic symptom items of the PHQ-9. Studies conducted in different patient populations, including people with systemic sclerosis (SSc), found either no significant differential item functioning (DIF) in somatic items of depression questionnaires or minimal DIF that did not significantly affect total questionnaire scores. It is possible that people with medical conditions who experience symptoms that may overlap with depression symptoms, including fatigue, changes in appetite, and sleep problems, do not report them on the PHQ-9 or PHQ-8 more than people without medical conditions due to a question ordering or context effect. The investigators will use the multinational Scleroderma Patient-centered Intervention Network (SPIN) Cohort to conduct a randomized experiment to examine whether awareness that depression symptoms are being assessed affects how people with a chronic illness report somatic symptoms of depression.
* OBJECTIVES The primary objective will be to evaluate differences in mean sum scores of PHQ-8 somatic items (sum of item 3 = sleep disturbances, item 4 = fatigue, and item 5 = changes in appetite) in people with SSc when the items are administered outside the context of a depression questionnaire compared to when they are administered in the context of a depression questionnaire. The secondary objective will be to evaluate differences in mean scores for each individual somatic symptom item.
* RECRUITMENT The SPIN Cohort is a large multinational cohort that collects longitudinal data on patient-reported outcomes from people living with SSc. It currently includes >1500 active participants recruited from 53 SPIN sites in Canada, the United States, Mexico, Australia, and France, Spain, and the United Kingdom. SPIN cohort participants are recruited during regular medical visits at SPIN recruitment sites, and written informed consent is obtained. Once enrolled in the Cohort, participants are sent an automated welcome email with instructions on how to activate their SPIN account and complete SPIN Cohort measures online. Cohort participants complete online assessments upon enrolment and at 3-month intervals. All SPIN Cohort participants who log in to the SPIN Cohort platform to complete a routine 3-month assessment will be included in this experiment.
* RANDOMIZATION The SPIN Cohort platform will be programmed to automatically randomize each participant via simple randomization in a 1:1 ratio to either the "Reordered items" arm or the "Original item order" arm.
* OUTCOMES The primary outcome variable will be the sum score of the 3 PHQ-8 somatic symptom item scores (item 3 = sleep disturbances, item 4 = fatigue, and item 5 = changes in appetite). The secondary outcome variables will be the individual item scores for items 3, 4, and 5.
* METHODS This is a two-arm parallel randomized controlled experiment. When SPIN Cohort participants log in to complete their routine assessment, they will be randomly assigned to complete either the standard PHQ-8 or a reordered version in which the 3 somatic symptom items (item 3 = sleep disturbances, item 4 = fatigue, and item 5 = changes in appetite) will be presented first, without any indication that they are part of a depression questionnaire, and the psychological symptom items will be presented later in the assessment protocol. Both primary and secondary analyses will be done as complete case analyses using between-groups t-tests.

ELIGIBILITY:
Inclusion Criteria:

* SPIN Cohort patients must have a systemic sclerosis (SSc) diagnosis based on 2013 American College of Rheumatology/European League Against Rheumatism criteria confirmed by a SPIN physician, be ≥18 years old, be able to give informed consent, and be fluent in English, French or Spanish.
* Participants must have access to a computer or tablet with internet access.

Exclusion Criteria:

* None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 851 (Actual)
Dates: Start 2025-01-17 (Actual); Primary Completion 2025-04-17 (Actual); Study Completion 2025-04-17 (Actual)

PRIMARY OUTCOMES:
Difference in mean sum PHQ-8 somatic item scores when administered outside and within a depression questionnaire context | At enrollment
  Scores obtained on the 8-item Patient Health Questionnaire (PHQ-8) range from 0 to 24, with higher scores indicating worse outcome. Individual items are scored on a 4-point scale ranging from 0 (not at all) to 3 (nearly every day). PHQ-8 somatic items will include items 3 (sleep problems), 4 (fatigue), and 5 (changes in appetite). The investigators will compare the mean sum score of somatic item scores between the "Reordered items" arm and the "Original item order" arm using a between-groups t-test.

SECONDARY OUTCOMES:
Difference in individual PHQ-8 somatic item mean scores when administered outside and within a depression questionnaire context | At enrollment
  Scores obtained on the 8-item Patient Health Questionnaire (PHQ-8) range from 0 to 24, with higher scores indicating worse outcome. Individual items are scored on a 4-point scale ranging from 0 (not at all) to 3 (nearly every day). PHQ-8 somatic items will include items 3 (sleep problems), 4 (fatigue), and 5 (changes in appetite). The investigators will compare mean scores of each individual item between the "Reordered items" arm and the "Original item order" arm using 3 between-groups t-tests.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Jewish General Hospital, Montreal, Quebec
  - Lady Davis Institute for Medical Research, Montreal, Quebec